CLINICAL TRIAL: NCT01911273
Title: A Phase 2, Randomized, Double Blind Study To Evaluate The Efficacy, Safety, Pharmacodynamics And Pharmacokinetics Of The Anti-alk-1 Monoclonal Antibody Pf-03446962 In Combination With Best Supportive Care Vs. Placebo Plus Best Supportive Care In Adult Patients With Advanced Hepatocellular Carcinoma Following Failure Of Sorafenib
Brief Title: A Study To Evaluate The Efficacy And Safety of The Investigational Drug PF-03446962 (A Monoclonal Antibody With Antiangiogenic Features) In Combination With Best Supportive Care Versus Placebo Plus Best Supportive Care In Patients Affected By Recurrent Liver Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8471005; 2013-001426-26 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular carcinoma; monoclonal antibody; ALK-1; best supportive care
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ascrinvacumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PF 03446962 plus best supportive care (BSC) (Experimental)
  Interventions: Drug: PF-03446962; Other: Best Supportive Care
- Placebo plus best supportive care (BSC) (Placebo Comparator): Placebo, IV, every 2 weeks, until disease progression, patient refusal or unacceptable toxicity, whichever occurs first
  Interventions: Other: Placebo; Other: Best Supportive Care

INTERVENTIONS:
Drug: PF-03446962 — PF 03446962 7 mg/kg, IV, every 2 weeks, until disease progression, patient refusal or unacceptable toxicity, whichever occurs first
  Arms: PF 03446962 plus best supportive care (BSC)
Other: Best Supportive Care — BSC may include medications and supportive measures deemed necessary to palliate disease related symptoms and improve quality of life
  Arms: PF 03446962 plus best supportive care (BSC)
Other: Placebo — Placebo will consist of Saline (0.9% w/v Sodium Chloride Injection, USP or NS)
  Arms: Placebo plus best supportive care (BSC)
Other: Best Supportive Care — BSC may include medications and supportive measures deemed necessary to palliate disease related symptoms and improve quality of life.
  Arms: Placebo plus best supportive care (BSC)

SUMMARY:
The primary purpose of the study is to explore whether treatment with PF-03446962 and best supportive care is better than placebo plus best supportive care in prolonging survival of patients affected by recurrent liver cancer. In addition, the study will explore if adding PF-03446962 to best supportive care is safe, how PF-03446962 is metabolized, if there are patients' characteristics (biomarkers) that may predict response to PF-03446962, and if PF-03446962 has any effect on the patients' quality of life.

DETAILED DESCRIPTION:
This study was terminated on June 24th, 2014 due to change in strategy of PF-03446962 clinical development. There were no safety or efficacy concerns regarding the study behind the decision to terminate the trial. The study was on temporary halt since March 10th and there are currently no patients on treatment or in the process of being randomized

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of locally advanced or metastatic liver cancer obtained by histology/cytology or by imaging
* Documented progression on or after treatment with sorafenib, confirmed by the Investigator upon review of appropriate imaging documentation
* Child Pugh Class A disease
* ECOG [Eastern Cooperative Oncology Group] Performance Status (PS) 0 or 1
* Mandatory tumor biopsy at study entry (pre-randomization, unless already collected after sorafenib progression but within 3 months of enrollment and no systemic anticancer therapies received)

Exclusion Criteria:

* Prior systemic treatment for advanced liver cancer other than sorafenib-including therapy
* Prior local therapy within 2 weeks of starting the study treatment
* Presence of main portal vein invasion by liver cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Kinki University Hospital, Department of Gastroenterology and Hepatology, Ōsaka-sayama, Osaka
  - National Cancer Center Hospital, Chuo-ku, Tokyo

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8471005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 3 participants were enrolled into this study as of termination date. One participant was assigned to receive PF-03446962 plus best supportive care (BSC) treatment and 2 participants were assigned to receive only BSC treatment.
Groups:
- PF-03446962 Plus BSC: PF-03446962 7 milligram per kilogram (mg/kg) was administered intravenously (IV) as 1-hour infusion every two weeks (q2w) plus BSC
- BSC Alone: BSC might vary depending on the participant's signs and symptoms, site current practice, and country practice and might include medications and supportive measures deemed necessary to palliate disease-related symptoms and improve quality of life.
Period: Overall Study
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Progression of Disease | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- PF-03446962 Plus BSC: PF-03446962 7 mg/kg was administered IV as 1-hour infusion q2w plus BSC
- Total: Total of all reporting groups
Arm/Group | PF-03446962 Plus BSC | BSC Alone | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Customized [Number; unit: Participants]
  18 to 44 Years | 1 (0.0) | 0 (NA) | 1
  45 to 64 Years | 0 (NA) | 2 (6.4) | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 2 | 2

OUTCOME MEASURES:

1. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time from first randomization to date of first documentation of objective tumor progression. If tumor progression data included more than (>) 1 date, the first date was to be used. TTP (in months) was calculated as first event date or last known progression-free date minus the first randomization date plus 1 divided by 30.4. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease per Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1).
Time Frame: Screening and every 8 weeks by calendar thereafter, up to 24 months after last participant randomization.
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 2
Months | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading

2. Primary Outcome: Overall Survival (OS)
Description: OS was the duration from date of randomization to date of death due to any cause. For participants who are alive, overall survival was censored at the last contact. Death was determined from adverse event (AE) data where outcome was death or from follow-up contact data where the participant current status was death.
Time Frame: From first randomization to date of death from any cause, whichever came first, assessed up to 24 months after last participant randomization
Population: Full analysis set (FAS) included all randomized participants regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 2
Months | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading

3. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time from randomization to first documentation of objective tumor progression or to death due to any cause, whichever occured first. If tumor progression data included >1 date, the first date was to be used. PFS (in months) was calculated as first event date minus first randomization date plus 1 divided by 30.4.
Time Frame: Screening and every 8 weeks by calendar thereafter, up to 24 months after last participant randomization.
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 2
Months | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading

4. Secondary Outcome: Objective Response Rate (ORR) - Percentage of Participants With Objective Response
Description: ORR was defined as the proportion of participants with confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.1, relative to all randomized participants. CR were those that persisted on repeat imaging study more than or equal to (>=) 4 weeks after initial documentation of response. PR was defined as >=30% decrease in the sum of diameters of target lesions and non CR/non PD to non-target lesions. Participants who did not have on study radiographic tumor re-evaluation or who died, progressed or dropped out for any reason prior to reaching a CR or PR were to be counted as non-responders in the assessment of ORR. A participant who initially met the criteria for a PR and then subsequently became a confirmed CR, was to be assigned a best response of CR.
Time Frame: Screening and every 8 weeks by calendar thereafter, up to 24 months after last participant randomization.
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Measure: Number; unit: Percentage of Participants
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 2
Percentage of Participants | NA — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading | NA — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading

5. Secondary Outcome: Duration of Response (DR)
Description: DR was defined as the time from the first documentation of objective tumor response to the first documentation of objective tumor progression or to death due to any cause, whichever occurred first. If tumor progression data included >1 date, the first date was to be used. DR (in months) was calculated as the end date for DR minus date of first CR or PR that was subsequently confirmed plus 1 divided by 30.4. CR was defined as disappearance of all target lesions and non-target, if any. PR was defined as >=30% decrease in the sum of diameters of target lesions and non CR/non PD to non-target lesions.
Time Frame: From first randomization to date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months after last participant randomization
Population: Subgroup of participants with objective response. Since objective response was not assessed in any of the participants, ideally the number of participants analyzed field should be 0 and the reason was insufficient data available to conduct adequate analysis due to premature termination of the study.
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants With Disease Control Rate (DCR) at 16 Weeks
Description: DCR was defined as the proportion of participants with confirmed CR or confirmed PR or a best response of stable disease (SD) >=16 weeks according to RECIST, relative to all randomized participants. CR was defined as disappearance of all target lesions. PR was defined as >=30% decrease in the sum of diameters of target lesions and non CR/non PD to non-target lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum diameters while on study.
Time Frame: as for outcome 5
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 2
Percentage of Participants | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading | NA [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading

7. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy-Hepatobiliary Questionnaire (FACT-Hep)
Description: Patient reported outcomes (PROs) were assessed using the FACT-Hep. The FACT-Hep included the FACT-general (FACT-G) and a hepatobiliary module, it consisted of the 27-item FACT-G, which assessed generic health-related quality of life (HRQoL) concerns, and the 18-item hepatobiliary subscale (HS), which assessed disease-specific issues. The questionnaire used a 5 point Likert scale from '0' "not at all" to '4' "very much" regarding how much each item was present in the last 7 days; lower score indicated severer symptom. Eight of the items (lack of energy, pain, weight loss, back pain, fatigue, stomach pain/discomfort, nausea, and jaundice) made up the Fact Hepatobiliary Symptom Index (FHSI 8) were considered to be symptoms specific to hepatobiliary cancer.
Time Frame: Screening, Cycle 1 Day1,8; Cycle >=2 Day1; End of treatment, survival follow-up up to 24 months after last participant randomization.
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 2
Units on scale | NA (NA) [NA to NA] — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading | NA (NA) — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading

8. Secondary Outcome: Maximum Serum Concentration (Cmax)
Time Frame: 1 hour (after start of infusion) on Day1 of Cycles 1, 2, 4, 6, and 8
Population: The pharmacokinetic (PK) concentration set consisted of all participants who were treated and had at least one concentration on at least 1 day of PK assessment.
Measure: Geometric Mean (Standard Error); unit: microgram per milliliter (mcg/mL)
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 0
microgram per milliliter (mcg/mL) | NA (NA) — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading |

9. Secondary Outcome: Trough Serum Concentration of PF-03446962 (Ctrough)
Time Frame: 0 hour (predose) on Day 1 of Cycles 1, 2, 4, 6, and 8
Population: The PK concentration set consisted of all participants who were treated and had at least one concentration on at least 1 day of PK assessment.
Measure: Geometric Mean (Standard Error); unit: mcg/mL
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 0
mcg/mL | NA (NA) — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading |

10. Secondary Outcome: Number of Participants With Human Anti-Human Antibodies (HAHA)
Time Frame: Cycle 1, 2, 4, 6, 8 Day 1 at 0 hour (pre-dose)
Population: The immunogenicity assessment consisted of all participants who had at least 1 sample on at least 1 day of immunogenicity assessment.
Measure: Number; unit: Participants
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 0
Participants | NA — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading |

11. Secondary Outcome: Presence of Sensitivity Signature
Description: Tumor molecular characteristics including but not limited to transcriptomic (RNA) signatures of sensitivity
Time Frame: Cycle 1 Day 1 (before infusion), Cycle 4 Day 1 (before infusion), at disease progression/participant withdrawal.
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Ratio to Baseline of Serum Circulating Protein Concentration
Description: Protein involved TGFB1, VEGF-A, VEGF-C, PIGF, Endoglin, BMP-9, VEGFR1, VEGFR2, VEGFr3, Ang-2, VEGF-D, CD54, CD106, and CCL2. Tumor molecular characteristics including but not limited to transcriptomic (ribonucleic acid) signatures of efficacy.
Time Frame: Cycle 1 Day 1 (before infusion), Cycle 4 Day 1 (before infusion), at disease progression/participant withdrawal.
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Measure: Number; unit: Percentage
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 0
Percentage | NA — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading |

13. Secondary Outcome: Observed Serum Concentration of Circulating Protein
Time Frame: Cycle 1 Day 1 (before infusion), Cycle 4 Day 1 (before infusion), at disease progression/participant withdrawal.
Population: FAS included all randomized participants regardless of what treatment, if any, was received.
Measure: Number; unit: mcg/mL
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Number analyzed (Participants) | 1 | 0
mcg/mL | NA — Due to the early termination of the study the incomplete data set was not reported because it would potentially skew the data, and is not statistically relevant, thus could be misleading |

ADVERSE EVENTS:
Time Frame: Day 1 up to 28 days after the last administration of study medication.
Description: Three participants were assigned to receive study treatment, as of study termination date. One participant was assigned to receive PF-03446962 plus BSC treatment and discontinued due to progression of disease; 2 were assigned to receive BSC only treatment and discontinued due to withdrawal of consent.
Arm/Group | PF-03446962 Plus BSC | BSC Alone
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PF-03446962 Plus BSC (N=1) | BSC Alone (N=2)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
This study was prematurely terminated due to a Sponsor decision not to pursue the clinical development of PF-03446962 as monotherapy in second-line hepatocellular carcinoma.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will provide manuscripts, abstracts, or the full text of any other intended disclosure (poster presentation, invited speaker or guest lecturer presentation, etc.) to Pfizer at least 30 days before they are submitted for publication or otherwise disclosed. If any patent action is required to protect intellectual property rights, Investigator agrees to delay the disclosure for a period not to exceed an additional 60 days.